CLINICAL TRIAL: NCT03341884
Title: A Phase 1, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics and Safety of Ipatasertib in Subjects With Mild, Moderate or Severe Hepatic Impairment Compared to Healthy Subjects
Brief Title: A Study of Ipatasertib in Participants With Mild, Moderate or Severe Hepatic Impairment Compared to Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP40200
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — ipatasertib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Normal Hepatic Function (Experimental): Participants with normal hepatic function will be administered a single oral dose of ipatasertib (100 mg).
  Interventions: Drug: Ipatasertib
- Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment (Child-Pugh Class A, score of 5 to 6, inclusive) will be administered a single dose of ipatasertib (100 mg).
  Interventions: Drug: Ipatasertib
- Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment (Child-Pugh Class B, score of 7 to 9, inclusive) will be administered a single dose of ipatasertib (100 mg).
  Interventions: Drug: Ipatasertib
- Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment (Child-Pugh Class C, score of 10 to 15, inclusive) will be administered a single dose of ipatasertib (100 mg).
  Interventions: Drug: Ipatasertib

INTERVENTIONS:
Drug: Ipatasertib — A single oral dose of 100 mg ipatasertib will be administered.
  Other Names: GDC-0068

SUMMARY:
This is a Phase 1 study evaluating the pharmacokinetics, tolerability and safety of a single dose of ipatasertib in participants with mild, moderate or severe hepatic impairment compared to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* In good health (except for specific inclusion criteria related to hepatic impairment), as determined by the Investigator, based on no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram, and vital signs
* Females will not be pregnant or breastfeeding, and must be either postmenopausal or agree to use a study-approved method of contraception from the time of signing the informed consent until 30 days after discharge
* Males will either be sterile or agree to use male condom with spermicide from check-in (Day -1) until 90 days following the dose of study drug

Additional Inclusion Criteria for Healthy Subjects Only:

- Liver enzyme tests must be less than or equal to the upper limits of normal

Additional Exclusion Criteria for Hepatic Impaired Subjects Only:

- Hepatic impairment must have a Child-Pugh score of 5 to 6 (mild), 7 to 9 (moderate), or 10 to 15 (severe) and have stable hepatic insufficiency within 1 month prior to Screening

Exclusion Criteria:

* History of ulcerative colitis or stomach or intestinal surgery or resection
* History of unstable diabetes mellitus
* History of alcoholism or drug addiction within 1 year prior to Check-in (Day -1)
* Use of oral, implantable, transdermal, or injectable contraceptives from the time of signing the informed consent (females only) or 10 days prior to Check-in through 45 days after the dose administration
* Poor peripheral venous access
* Receipt of blood products within 2 months prior to check-in

Additional Exclusion Criteria for Healthy Subjects Only:

* Use of any tobacco- or nicotine-containing products within 6 months prior to check-in and during the entire study
* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder

Additional Exclusion Criteria for Hepatic Impaired Subjects Only:

* Any evidence of progressive liver disease that has worsened or is worsening within 1 month prior to the screening visit
* Participant has shown evidence of hepatorenal syndrome
* Ascites requiring paracentesis
* Participant has required treatment for GI bleeding within 12 months prior to Check-in
* Participant has required additional medication for hepatic encephalopathy within the 12 months (6 months for severe hepatic impairment) prior to check-in
* Total bilirubin levels >6 mg/dL

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve (AUC) from 0 to Infinity (AUC0-inf) of Ipatasertib | up to Day 15
  AUC0-inf is defined as AUC extrapolated from Hour 0 to infinity of ipatasertib in the plasma.
Maximum Observed Plasma Concentration (Cmax) of Ipatasertib | up to Day 15
  Maximum observed concentration of ipatasertib as determined by measuring drug concentration in blood samples over time.

SECONDARY OUTCOMES:
Percentage of Participants with Treatment-Emergent Adverse Events (AE) | up to Day 15
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time to Reach Maximum Observed Concentration (tmax) of Ipatasertib | up to Day 15
  Time from dose administration to observed maximum serum concentration for ipatasertib as determined by measuring drug concentration in blood samples over time.
AUC from 0 to last measurable concentration (AUC0-t) | up to Day 15
  Area under the plasma concentration-time curve from Hour 0 to the last measurable concentration of ipatasertib.
Half-life (t1/2) of Ipatasertib | up to Day 15
  Half-life of ipatasertib is the time elapsed for the drug concentration to decrease by half as determined by measuring drug concentration in blood samples over time.
Apparent Plasma Clearance (CL/F) of Ipatasertib | Up to Day 15
  Apparent clearance (CL/F) of ipatasertib, where CL is clearance and F is bioavailability (relative amount of extravascularly-administered drug that reaches systemic circulation unchanged). Determined by measuring drug concentration in blood samples over time.
Apparent Volume of Distribution (V/F) of Ipatasertib | up to Day 15
  Apparent volume of distribution (V/F) during the terminal phase of ipatasertib.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, Inc., Miami, Florida
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - American Research Corporation Inc., San Antonio, Texas